CLINICAL TRIAL: NCT03898427
Title: Quantification of Improvement in Scratch Behavior and Sleep in Patients With Atopic Dermatitis on Standard of Care Treatment
Brief Title: Scratch Behavior Under Standard of Care
Acronym: SOC
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Other Study IDs: H-38472
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Atopic Dermatitis
Keywords: Wearable devices; Scratch; Sleep
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with atopic dermatitis: Sensor technology and digital measures will be used to evaluate scratch and sleep in individuals with atopic dermatitis receiving standard of care treatments (SOC) who will wear watch-like wrist actigraphy devices, sleep monitor, polysomnography, and videography.
  Interventions: Device: Wrist Actigraphy Devices; Device: Polysomnography; Device: Videography

INTERVENTIONS:
Device: Wrist Actigraphy Devices — A watch-like wearable sensor
  Other Names: GENEActiv Watch
Device: Polysomnography — Sleep Monitor
Device: Videography — Thermal Camera

SUMMARY:
Wrist-worn accelerometers and associated data analysis platforms will provide quantitative and qualitative knowledge regarding the action of scratching and sleep quantity in a symptomatic Atopic Dermatitis (AD) population. The overall research aim is to evaluate the sensitivity of digital devices to capture drug-induced (standard of care treatments; SOC) quantitative changes in nighttime scratch and sleep quantity in AD subjects. In the current study, the investigators aim to evaluate the ability of wrist-worn accelerometers to detect significant and clinically meaningful changes in scratch behavior and sleep quantity in patients with symptomatic AD aged 2 to 75 years, receiving topical SOC treatment for AD. To evaluate this experimental paradigm, using wearable accelerometers, traditional patient-reported outcome measures/observer-reported outcome (ObsRO) (PRO/ObsRO), thermal videography and physician assessments of AD will be assessed in a well-controlled observational methodology study that has both an in-patient and out-patient portions within the study.

DETAILED DESCRIPTION:
This open label study is to evaluate the ability of a wrist-worn accelerometry device to detect scratch and sleep quantity changes in patients with Atopic Dermatitis (AD) receiving Standard of Care (SOC) treatment. Subjects, age 2 to 75 years, with symptomatic AD will be recruited.

The study will be comprised of an initial screening/baseline clinic visit when subject will be diagnosed with symptomatic AD, screened and enrolled in the study after signing an informed consent (or parents/guardians and assent when appropriate). The subject will start or modify a SOC treatment course at the physician's discretion, and thereafter will be followed up for a total of 2 weeks for the purposes of the study. During those 2 weeks, the subject will wear two wrist worn accelerometry devices. The subject will also have to complete daily PRO/ObsRO related to itch, sleeping habits, quality of life, and device comfort questionnaires (parent/guardian will complete as appropriate) and may also participate in an optional daily photography taken of a single lesion (optional and for adult subjects only 18-75 years of age). The subject will also be asked to come and stay overnight at the sleep clinic for an overnight between Days 1-3, for thermal video recording overnight. An optional additional night (immediately following the first clinic overnight; between days 2-4) with video and polysomnography (PSG) may occur (subjects must be 18-75 years of age to participate in this aspect of the study). The subjects will be asked to return to the clinic on days 8 and 15 for clinician-based assessments. At the completion of the study, Day 15 (+3 day) the subjects will return the devices, and will complete PRO/ObsRO questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged between ≥2 years of age and <75 years of age at Day 1.
2. Written informed consent from subject/parent(s)/guardian(s) and assent from the subject, where assent is applicable (for those subjects under 18 years of age).
3. Subject and parent(s)/guardian(s) are willing and able to comply with study instructions, study visits, and procedures.
4. Native English speakers or demonstrated fluency in English (both subject and parent(s)/guardian(s) in the case of minors).
5. Have a clinical diagnosis of AD according to the criteria of Hanifin and Rajka.

Exclusion Criteria:

1. Has any clinically significant medical disorder, condition, disease (including active or potentially recurrent non AD dermatological conditions and known genetic dermatological conditions that overlap with AD, such as Netherton syndrome) or clinically significant finding at screening that precludes subject's participation in study activities.
2. Allergy to polyurethane resin (strap/wristband component), skin nickel allergy, silicone, and/or adhesives.
3. Has documented non-AD related insomnia, sleep apnea or other sleep-related disorders (e.g., narcolepsy, restless legs syndrome, circadian rhythm disorder).
4. Has unstable AD (Total BSA>40%) (including a significant active systemic or localized infection).

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with atopic dermatitis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Quantification of scratch using GENEActiv watches to assess triaxial accelerometry following standard of care (SOC) treatments | From enrollment through the end of visit 5 (15 days +/- 3 days).
  One GENEActiv watch will be used on each hand at a sampling rate of 100 Hz to measure movement in the x, y, and z direction. The movement will be analyzed using the algorithm described by Cole et al. to differentiate between periods of wakefulness and sleep following SOC treatments.
Quantification of sleep using polysomnography following SOC treatment | From enrollment through the end of visit 5 (15 days +/- 3 days).
  Polysomnography (PSG) will be used to report the number of sleep occurrences and appropriate sleep staging following SOC treatments based on the scoring guide provided by the American Academy of Sleep Medicine (AASM). The following sleep stages will be scored: Stage W (wakefulness), Stage N1 (NREM 1), Stage N2 (NREM 2), Stage N3 (NREM 3), Stage N (NREM), and Stage R (REM).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Thomas, PhD, MBA, Principal Investigator — Boston University, Department of Anatomy and Neurobiology
Locations (1):
- Evans Biomedical Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No